CLINICAL TRIAL: NCT03411226
Title: Management of Recurrent Inguinal Hernia After Previous Open Preperitoneal Repair: Is Re-TREPP Feasible?
Brief Title: Feasibility of Re-TREPP in Patients With a Recurrent Inguinal Hernia After Previous TREPP Repair
Acronym: re-TREPP
Status: Completed | Type: Observational
Sponsor: Alexandra Persoon (Other)
Responsible Party: Sponsor-Investigator, Alexandra Persoon, Drs. A.M. Persoon, St Jansdal Hospital
Organization: St Jansdal Hospital (Other)
Other Study IDs: 01012006
Record Dates: First submitted 2018-01-04; First posted 2018-01-26 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Recurrent Inguinal Hernia
Keywords: Inguinal Hernia; TREPP; Recurrence
MeSH Terms: conditions — Hernia, Inguinal; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- re-TREPP: Patients who presented with a recurrent inguinal hernia after previous TREPP repair.
  Interventions: Procedure: re-TREPP

INTERVENTIONS:
Procedure: re-TREPP — repeated hernia repair via the TREPP technique

SUMMARY:
The Trans REctussheath PrePeritoneal (TREPP) mesh repair was introduced in 2006 to decrease the risk of postoperative inguinal pain in hernia surgery. For the repair of a recurrent inguinal hernia after a primary TREPP an alternative open anterior route (Lichtenstein) may seem the most logical option, but coincides with an increased risk of chronic postoperative inguinal pain. Therefore, this study aimed to evaluate the feasibility of a second TREPP procedure to repair a recurrent inguinal hernia after an initial TREPP repair. The hypothesis was that the technique is possible and does not lead to an increased risk of postoperative pain.

DETAILED DESCRIPTION:
Since the development and introduction of TREPP in 2006, TREPP has been the standard operation technique for all patients who present in St. Jansdal Hospital with an inguinal hernia. The electronic patient files of all consecutive patients who were operated at the St Jansdal hospital via TREPP between January 2006 and December 2013 were retrospectively investigated. This patient list was retrieved by an electronic search using the assigned operation codes. Adult patients who had developed a recurrent inguinal hernia and had undergone a re-TREPP were included in this study. A case report form was filled in for each patient that underwent a re-TREPP. Baseline data such as operation time, Body Mass Index (BMI), operation technique, number of conversions, aetiology of the recurrence, type of anesthesia and American Society of Anesthesiology (ASA) classification were retrospectively reviewed through patient files and operation reports. Co-morbidities were extracted from the files. Information on short term complications was taken from the notes of telephone consultation 2 and 30 days postoperatively, which is the local standard protocol for follow-up. Patients were invited for a long-term follow-up (>30 days postoperative) at the outpatient department for physical examination, or they were visited at home by the investigator. Written informed consent was obtained from all patients who were included for a long term follow-up. A case report form was used for each patient, in order to standardize the investigation. All patients were asked if they experienced any pain or discomfort. If there was pain, the Visual Analogue Scale and Pain Disability Index questionnaire were filled in. All patients were asked if sexual complaints occurred since the operation. Written informed consent was obtained from all patients who were clinically evaluated. Recurrent inguinal hernia was defined as a reappearance of the inguinal hernia, diagnosed by physical examination (a reducible bulge with positive Valsalva).

This was a retrospective case series. Since the numbers were small, no statistical analysis was performed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who had developed a recurrent inguinal hernia and had undergone a re-TREPP.

Exclusion Criteria:

* Children (age <18 years)
* Exclusion criterium for long term follow up: no informed consent obtained.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: From all re-TREPP patients (n=19), the mean age at time of the re-operation was 68 years (range 56-86 years). All included patients, 18 males and 1 female, were classified with the American Society of Anesthesiologists (ASA) classification ≤3.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2015-11-27 (Actual); Primary Completion 2015-12-10 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
Chronic postoperative inguinal pain according to Visual Analogue Scale. | This was assessed between >30 days postoperative and the moment of evaluation (up to 95 months postoperative).
  All patients who reported chronic pain (>30 days postoperative) were asked to fill out the Visual Analogue Scale. This was a horizontal line of 100 millimeters long. Patients were asked to mark the point that indicated the amount of pain that they experienced. The length between the left anchor 'no pain' and the patients mark was measured, providing a range of 0 to 100. A greater score indicated greater pain intensity.
Chronic postoperative pain according to Pain Disability Index | This was assessed between >30 days postoperative and the moment of evaluation (up to 95 months postoperative).
  All patients who reported chronic pain (>30 days postoperative) were asked to fill out the Pain Disability Index questionnaire.

SECONDARY OUTCOMES:
Re-recurrence rate | This was assessed by reviewing the electronic patient files and via a physical examination at the long term follow-up (ranging from >30 days postoperative, up to 95 months postoperative).
  The number of second recurrences after re-TREPP repair
Short term complications | Complications occuring from the start of the operation up to 30 days postoperative.
  Short term complications included: hematoma, wound infection, re-admission rate, medical complications and death. These complications were retrospectively analyzed via the electronic patient files.
Sexual complaints related to re-TREPP | This was assessed between >30 days postoperative and the moment of evaluation (up to 95 months postoperative).
  All patients were asked if they experienced any sexual problems related to the re-TREPP surgery. The question was answered with 'yes', 'no' or 'not sure'.

CONTACTS AND LOCATIONS:
Overall Officials: Giel G Koning, MSc, PhD, Study Chair — St Jansdal Hospital

IPD SHARING:
Plan to Share IPD: No